CLINICAL TRIAL: NCT02344186
Title: Effects of Liraglutide on Endoplasmic (ER) Stress in Obese Patients With Type 2 Diabetes
Brief Title: Effects of Liraglutide on ER Stress in Obese Patients With Type 2 Diabetes
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Temple University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 21440
Record Dates: First submitted 2015-01-14; First posted 2015-01-22 (Estimated); Last update posted 2022-07-29 (Actual); Status verified 2022-07

CONDITIONS: Type 2 Diabetes
Keywords: diabetes, ER stress, glucagon-like peptide-1 analogs
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Liraglutide

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Liraglutide (Experimental): Liraglutide will be started first with 0.6 mg/d for 1 week, then increased to 1.2 mg/d from week 2 to week 12, followed by 1.8 mg/d from week 12 to week 24.
  Interventions: Drug: Liraglutide
- Placebo (Placebo Comparator): Subjects will receive placebo for 12 weeks.
  Interventions: Drug: Liraglutide

INTERVENTIONS:
Drug: Liraglutide — Crossover design - 24 weeks on active drug and 12 weeks daily placebo
  Other Names: Victoza

SUMMARY:
The main objective of the study will be to test the hypothesis that treatment with Liraglutide will decrease ER stress and adipose tissue in obese patients with type 2 diabetes. Experimental Approach: The investigators will use a prospective, single blind, placebo controlled study design to study 12 obese patients with type 2 diabetes mellitus (T2DM). 6 patients will first receive Liraglutide for 24 weeks followed by placebo for 12 weeks. The other 6 patients will first receive placebo for 12 weeks followed by Liraglutide for 24 weeks.

Measurements: The investigators will determine glycemic control (with HbA1c), body composition (bioelectric impedance analysis), insulin sensitivity (with hyperinsulinemic-euglycemic clamps), insulin secretion (with oral glucose tolerance testing), energy balance (calories in vs. calories out), plasma lipid levels and obtain subcutaneous fat biopsies to determine ER stress response markers before and after placebo and before and after Liraglutide treatment.

DETAILED DESCRIPTION:
This will be a prospective, single-blind, placebo-controlled study with a crossover design.

Visit Procedures: After a 1 month run-in period during which there will be no changes in medications, physical activity or diet, patients will be randomly divided into 2 groups of 6 patients each. Subjects have a 50:50 chance of being randomized to either group 1 or group 2.

In Group 1, (n=6), liraglutide will be started first with 0.6 mg/d for 1 week, then increased to 1.2 mg/d from week 2 to week 12, followed by 1.8 mg/d from week 12 to week 24. Group 1 patients will then be switched from liraglutide to placebo injections for another 12 weeks. For subjects in Group 1 the placebo period (weeks 24 to 36 will be the washout period.

Group 2 patients (n=6) will be started with placebo for 12 weeks and then switched to liraglutide for the next 24 weeks (0.6 mg/d for 1 week, 1.2 mg/d for 11 weeks and 1.8 mg/d for 12 weeks).

Assessment of Efficacy

Outpatient visits:

During the entire study, all patients (Groups 1 and 2) will perform home glucose monitoring 7 times/day (pre and ~ 2 h post breakfast, lunch and dinner and bedtime) and will be seen at Temple University Hospital as outpatients at 4 week intervals.

One week before the first, second or third and final inpatient visit, patients will undergo a 75, gram 2-hour oral glucose tolerance test.

Inpatient visits:

All patients (Groups 1 and 2) will be studied in our Clinical Research Center (CRC) at Temple University Hospital in the morning after an overnight fast, at the end of the run-in period (Week 0 ) and again at Weeks 12, 24 and 36. All study patients will be admitted to the CRC the evening before their study and discharged in the afternoon of the following day.

During the inpatient visits, the following procedures will be performed.

1. At baseline and again at weeks 12 and 36, subcutaneous fat biopsies will be obtained from the lateral aspect of one thigh by a surgeon as described (8) for determination of ER stress markers. In brief, the skin will be cleaned with betadine and anesthetized with 1% lidocaine without epinephrine in a field block pattern (at 2 X 3 in). (We have found that injection of lidocaine too close to the biopsy site interfered with the measurement of acetyl-CoA). After an incision (~ 1 in.) will be made through the skin, ~ 300 mg of fat will be mobilized and excised. The fat will be dropped immediately into isopentane, kept at its freezing point (-160°C) by liquid nitrogen. The frozen fat will be stored at -70°. To screen for changes in unfolded protein response (UPR) genes, we will first perform an UPR PCR microarray (SA Biosciences, Frederick, MD) using pooled fat biopsy extracts. This array profiles expression of 84 key genes recognizing and responding to misfolded protein accumulation in the ER. Significant changes (> 1.5 fold comparing post vs. pre drug biopsies) will then be confirmed by real time reverse transcription (RT)-PCR of the UPR messenger RNAs (mRNAs). Thus, mRNAs of the identified UPR markers (for instance, GRP78, X-box-binding-protein 1 (XBP-1), activating transcription factor 4 (ATF4), activating transcription factor 6 (ATF6), protein disulfide isomerase (PDI), calreticulin, calnexin) will be measured by real time RT-PCR in triplicate and normalized against 18s and β-actin mRNAs and will be expressed as arbitrary units. The respective proteins will be analyzed by Western blots.
2. Glycemic control will be assessed by

   1. measurement of HbA1c
   2. patients home glucose monitoring records
3. Determination of insulin resistance will be determined (with euglycemic-hyperinsulinemic clamping with use of stable isotopes for determination of peripheral (GRd) and hepatic (GRa) insulin action as described (18).
4. . Determination of energy balance, which will be calculated as change in fat mass (by bioelectric impedance analysis) plus total energy expenditure (determined with indirect calorimetry and the doubly labeled water method) (17).
5. Postabsorptive blood samples will be obtained for determination of plasma lipids (total cholesterol, LDL, HDL and triglycerides).
6. Assessment of changes in insulin secretion will be determined with Oral Glucose Tolerance Testing.

ELIGIBILITY:
Inclusion Criteria:

* Patients with established type 2 diabetes, BMI 27-35, Age - 18-75 years, HbA1c 7-10%, patients treated with exercise, diet, metformin and/or alpha glucosidase inhibitors (all up to ½ of their maximal dose) or pioglitazone (up to 30 mg/d), ability to provide informed consent before any trial-related activities.

Exclusion Criteria:

* Patients with pancreatitis or a history of pancreatitis, patients with HbA1c < 7% or > 10%, type 2 diabetic patients treated with insulin, sulfonylureas, meglitinides, dipeptidyl peptidase-4 (DPP4) inhibitors, glucagon-like peptide-1 (GLP1) agonists or corticosteroids, patients with hypoglycemia unawareness and with impaired liver functions (≥ 2.5 times the upper normal limit), known or suspected allergy against liraglutide or contraindications to liraglutide (as specified in the product prescribing information), pregnancies, breastfeeding or intention of becoming pregnant or not using adequate contraceptive measures, patients with a personal or family history of medullary thyroid cancer and patients with Multiple Endocrine Neoplasia type 2.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2014-05; Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in unfolded protein response markers | baseline, 6 months, 9 months
  Changes in unfolded protein response markers in adipose tissue biopsy samples. Specifically, the investigators will determine changes in mRNA (by RT-PCR) and protein (by Western blots) levels of the following ER stress markers: GRP78, ATF4, XBP-1s, PDI, calreticulin and calnexin.

SECONDARY OUTCOMES:
Insulin sensitivity | baseline, 3 months, 6 months and 9 months
  Changes in insulin resistance will be determined by measuring changes in total body glucose uptake and in plasma free fatty acid (FFA) levels during euglycemic-hyperinsulinemic clamping.
Glucose control | baseline, 1 month, 2 months, 3 months, 4 months, 5 months, 6 months, 7 months, 8 months, 9 months
  Glucose control will be assessed by monthly A1c determinations.
Energy expenditure | baseline, 3 months, 6 months, 9 months
  Changes in energy expenditure will be assessed by indirect calorimetry
Body weight | baseline, 1 month, 2 months, 3 months, 4 months, 5 months, 6 months, 7 months, 8 months, 9 months
  Patients will be weighed monthly
Body composition | baseline, 3 months, 6 months and 9 months
  Body composition will be determined using bioelectrical impedance.
Beta cell function | baseline, 6 months, 9 months
  Subjects will undergo an oral glucose tolerance tests(OGTT) to assess beta cell function.

CONTACTS AND LOCATIONS:
Overall Officials: Ajaykumar D Rao, MD, Principal Investigator — Temple University
Locations (1):
- Temple University Hospital, Philadelphia, Pennsylvania, United States